CLINICAL TRIAL: NCT01485029
Title: Streptococcus Pneumoniae Nasopharyngeal Carriage Among Children Attending Day-care Centres in the Alpes Maritimes. Substudy: Enterobacterial Intestinal Carriage and Susceptibility to 3rd Generation Cephalosporins
Brief Title: Streptococcus Pneumoniae Nasopharyngeal Carriage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Department of Clinical Research and Innovation (Other)
Responsible Party: Sponsor-Investigator, Department of Clinical Research and Innovation, Pr PRADIER, Centre Hospitalier Universitaire de Nice
Organization: Centre Hospitalier Universitaire de Nice (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 11-APN-01
Record Dates: First submitted 2011-09-23; First posted 2011-12-05 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2011-12

CONDITIONS: Nursery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NP children (Experimental): Nasopharyngeal (NP) aspirate with a small flexible canule to obtain NP swabs
  Interventions: Procedure: Nasopharyngeal (NP) aspirate

INTERVENTIONS:
Procedure: Nasopharyngeal (NP) aspirate — Nasopharyngeal (NP) aspirate with a small flexible canule to obtain NP swabs

SUMMARY:
Antibiotic consumption and antimicrobial resistance remain notoriously high in France, particularly among children below three years of age. In France, the pneumococcal conjugate vaccine was officially recommended for all children under two in 2003, and consequently changes occurred in Streptococcus pneumoniae serotype distribution. Bacterial carriage among children attending day-care centres may result from vaccine- and antibiotic-driven selective pressure with possible repercussions on the community.

DETAILED DESCRIPTION:
Antibiotic consumption and antimicrobial resistance remain notoriously high in France, particularly among children below three years of age. In France, the pneumococcal conjugate vaccine was officially recommended for all children under two in 2003, and consequently changes occurred in Streptococcus pneumoniae serotype distribution. Bacterial carriage among children attending day-care centres may result from vaccine- and antibiotic-driven selective pressure with possible repercussions on the community.

To identify prevalence (rates) and trends in antibiotic resistance patterns in Streptococcus pneumoniae (SP) among children attending day-care centres, as well as antibiotic prescriptions and vaccine rates, nasopharyngeal (NP) carriage was monitored, by conducting five cross-sectional surveys from January to March 1999, 2002, 2004, 2006 and 2008 among these children in the area of the Alpes Maritimes, in South-Eastern France.

Interventions promoting prudent antibiotic use (PAU) took place in 2000 and since 2003, with temporary effectiveness but national prescription rates are reported to be currently increasing again. A new pneumococcal conjugate vaccine covering more serotypes (13-valent) now replaces the previous one. In this situation, a new cross-sectional survey in day-care centres with the same design may answer the following questions.

* Increasing antibiotic susceptibility was observed during past successive surveys. Has this trend been sustained to this day?
* Are antibiotics prescription rates among children attending day-care centres still decreasing, have they stabilized, or are they on the rise again reflecting recently reported national trends?
* Regarding choice of antimicrobial treatment, are 3rd generation cephalosporin increasingly prescribed rather than aminopenicillins?
* Is implementation of the new wider spectrum pneumococcal conjugate vaccine exerting changes on serotype distribution and thus on the nasopharyngeal ecosystem of these children? These parameters will be useful to renew, or even reinforce, and adapt professional guidelines and community-oriented messages concerning prudent antibiotic use.

Sub-study: Antibiotic-resistant enterobacteriaceae, initially observed in the hospital setting, are currently spreading within the community, especially extended-spectrum beta-lactamase-producing enterobacteriaceae, threatening antibiotic effectiveness in case of infection. Such infections with Enterobacteriaceae, in particular urinary tract infections, can occur among children. Prevalence rates of such carriage among children attending day-care centres is unknown, although they are highly exposed to antibiotics in relation with frequent respiratory tract infections, in particular to 3rd generation cephalosporins. To assess this prevalence rate, faecal samples from children attending day-care centres will be collected during the cross-sectional nasopharyngeal survey quoted above.

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 3 months to 4 years
* Attending a day care center
* Parents give informed consent

Exclusion Criteria:

* parents refusal

Ages: 3 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Streptococcus pneumoniae nasopharyngeal carriage among children attending day-care centres, and Streptococcus pneumoniae antibiotic susceptibility Substudy: Enterobacterial intestinal carriage and susceptibility to 3rd generation cephalosporins | one day

SECONDARY OUTCOMES:
•Antibiotics prescriptions within the 3 previous months in children's health booklets and in a questionnaire completed by parents | one day
• Immunization status for pneumococcal conjugate vaccine PCV7-type vaccine from children's health books and from day care centres health files | one day
• Pneumococcal serotypes distribution compared to immunization status | one day
• Comparison of the data above with the previous five cross-sectional surveys | one day

CONTACTS AND LOCATIONS:
Overall Officials: Christian PRADIER, PU-PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Hôpital Archet 1, Nice, France